CLINICAL TRIAL: NCT04628403
Title: Effects of Clinical Interventions for the Management of Late Start Muscular Pain (Doms) in the Post-exercise Recovery Process
Brief Title: Effects of Clinical Interventions for the Management of Late Start
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: São Paulo State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIRIO_STUDY
Record Dates: First submitted 2020-10-26; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Athletes
Keywords: Lasertherapy; Shockwaves; Massage; Sports Medicine; Athletic Performance
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the results assessor will not be aware of the subject allocation group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (No Intervention)
- shock waves (Experimental)
  Interventions: Device: shock waves
- massage (Experimental)
  Interventions: Other: massage
- lasertherapy (Experimental)
  Interventions: Device: lasertherapy

INTERVENTIONS:
Other: massage — clinical interventions, of mechanophysiological origin for the treatment of symptoms corresponding to DOMS, after exercise
  Arms: massage
Device: lasertherapy — lasertherapy
  Arms: lasertherapy
Device: shock waves — shock waves
  Arms: shock waves

SUMMARY:
Introduction: Late-onset muscle pain (DOMS) is characterized by a type of temporary muscle damage, common after high-intensity exercise. In addition to pain, DOMS clinically generates muscle stiffness, reduced joint range of motion, muscle weakness and reduced peak torque. In this regard, in order to accelerate the recovery of body systems and treat symptoms of DOMS, the management of different types of interventions has been observed, supporting the clinical practice, based on evidence. Objectives: To investigate the effect of different types of clinical interventions for the treatment of DOMS. Material and methods: For the clinical trial, 50 ultramarathon and rowing athletes of both sexes, aged between 18 and 60 years old, will be recruited randomly into four possible groups: control (CG), shock waves (G1) , massage (G2) and laser therapy (G3). The evaluation moments will be as follows: minutes before exercise (M1); immediately after exercise (M2); immediately after applying the recovery technique (M3); and 24 hours after exercise (M4) and the evaluated outcomes will be: pain, psychological aspects, functional test and blood markers.

ELIGIBILITY:
Inclusion Criteria:

* Professional athletes;
* Age over 18 years;
* Both sexes;
* Not having recent injuries

Exclusion Criteria:

* Participants who do not complete all the proposed collection moments
* who do not agree to participate will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2021-01-29 (Estimated); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
PAIN | 7 days
  pain systemic and located in quadriceps, assessed using a visual analog scale (0-10), with 0 indicating no pain and 10 the worst possible pain
SATISFACTION | 7 days
  Brunel's Mood Scale (BRUMS), with ratings from 0 to 4 where, 0 represents nothing; 1 represents a little, 2 indicates moderately; 3 reports a lot; and 4 corresponds to extremely

SECONDARY OUTCOMES:
MUSCLE STRENGTH | 7 days
  measured through a functional test entitled sit and stand. It is a test initially developed by researchers at UFRJ that consists of asking the subject to try to sit and stand in sequence, with the guidance of not using any support, for example the help of the hands or knees to obtain additional balance, leaving thus, that the musculature alone performs the function recruited

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Estado do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided